CLINICAL TRIAL: NCT00196404
Title: A Multicenter, Randomized, Double-blind Study to Evaluate the Safety and Efficacy of DR-3001 Versus Placebo in Women With Overactive Bladder
Brief Title: Study to Evaluate the Safety and Efficacy of DR-3001 Versus Placebo in Women With Overactive Bladder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duramed Research (Industry)
Responsible Party: Duramed Protocol Chair, Duramed Research, Inc
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BR-OXY-202
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Urinary Incontinence
Keywords: overactive bladder; urge incontinence; urinary incontinence
MeSH Terms: conditions — Urinary Incontinence; Urinary Bladder, Overactive; Urinary Incontinence, Urge

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: DR-3001a
- 2 (Experimental)
  Interventions: Drug: DR-3001b
- 3 (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: DR-3001a — 4mg daily vaginally
  Arms: 1
Drug: DR-3001b — 6 mg vaginally daily
  Arms: 2
Other: Placebo — Administered vaginally to match experimental arms
  Arms: 3

SUMMARY:
This is a placebo-controlled, double-blind study to evaluate the safety and efficacy of two doses of DR-3001 in women with overactive bladder who have symptoms of predominant or pure urge incontinence, urinary urgency and elevated urinary frequency

DETAILED DESCRIPTION:
This is a multi-center, randomized, placebo-controlled study to compare two doses of DR-3001 to placebo for a 12-week treatment period. The overall duration of patient participation will be for approximately 19 weeks. Patients will be required to keep a daily diary record of study medication use and incontinence episodes

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of overactive bladder and incontinence for at least 6 months
* Using birth control or menopausal
* Willing to discontinue current medication for overactive bladder

Exclusion Criteria:

* Pregnant or given birth in the last 6 months
* Three or more urinary tract infections a year
* Uncontrolled glaucoma, hypertension, diabetes or myasthenia gravis
* History of bladder cancer, ulcerative colitis or severe constipation
* Any contraindication to vaginal delivery systems

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2004-10; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Change in the total weekly number of incontinence episodes | Baseline to Treatment Week 12/Premature Discontinuation

SECONDARY OUTCOMES:
Average daily urinary frequency | Baseline to Treatment Week 12/Premature Discontinuation
Proportion of patients with no incontinence episodes | Baseline to Treatment Week 12/Premature Discontinuation
Average void volume | Baseline to Treatment Week 12/Premature Discontinuation
Average severity of urgency | Baseline to Treatment Week 12/Premature Discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Principal Investigator — Duramed Research
Locations (48):
- United States (46):
  - Duramed Investigational Site, Birmingham, Alabama
  - Duramed Investigational Site, Huntsville, Alabama
  - Duramed Investigational Site, Mobile, Alabama
  - Duramed Research Site, Phoenix, Arizona
  - Duramed Research Site, Tucson, Arizona
  - Duramed Investigational Site, Little Rock, Arkansas
  - Duramed Investigational Site, San Diego, California
  - Duremed Research Site, San Diego, California
  - Duramed Investigational Site, Aurora, Colorado
  - Duramed Research Site, Colorado Springs, Colorado
  - Duramed Investigational Site, Denver, Colorado
  - Duramed Investigational Site, Waterbury, Connecticut
  - Duramed Investigational Site, Aventura, Florida
  - Duramed Research Site, Gainesville, Florida
  - Duramed Investigational Site, Decatur, Georgia
  - Duramed Research Site, Sandy Springs, Georgia
  - Duramed Investigational Site, Boise, Idaho
  - Duramed Investigational Site, Boise, Indiana
  - Duramed Investigational Site, Evansville, Indiana
  - Duramed Investigational Site, Fort Wayne, Indiana
  - Duramed Investigational Site, Indianapolis, Indiana
  - Duramed Investigational Site, Jeffersonville, Indiana
  - Duramed Investigational Site, Meridian, Indiana
  - Duramed Investigational Site, Shreveport, Louisiana
  - Duramed Investigational Site, Jackson, Mississippi
  - Duramed Investigational Site, Lebanon, New Hampshire
  - Duramed Investigational Site, Edison, New Jersey
  - Duramed Investigational Site, Livingston, New Jersey
  - Duramed Investigational Site, Moorestown, New Jersey
  - Duramed Investigational Site, Williamsville, New York
  - Duramed Investigational Site, Portland, Oregon
  - Duramed Investigational Site, Lancaster, Pennsylvania
  - Duramed Investigational Site, Philadelphia, Pennsylvania
  - Duramed Investigational Site, Providence, Rhode Island
  - Duramed Investigational Site, Charleston, South Carolina
  - Duramed Investigational Site, Jackson, Tennessee
  - Duramed Investigational Site, Memphis, Tennessee
  - Duramed Investigational Site, Nashville, Tennessee
  - Duramed Investigational Site, Dallas, Texas
  - Duramed Research Site, Houston, Texas
  - Duramed Investigational Site, San Antonio, Texas
  - Duramed Research Site, Waco, Texas
  - Duramed Investigational Site, Salt Lake City, Utah
  - Duramed Investigational Site, Seattle, Washington
  - Duramed Research Site, Tacoma, Washington
  - Duramed Investigational Site, Milwaukee, Wisconsin
- Canada (2):
  - Duramed Investigational Site, Vancouver, British Columbia
  - Duramed Investigational Site, Toronto, Ontario

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- See also: MedLine Plus - Urinary Incontinence — http://www.nlm.nih.gov/medlineplus/urinaryincontinence.html